CLINICAL TRIAL: NCT00526942
Title: Computer-Based Cognitive Training in Normal Healthy Aging: Pilot Study of Behavioral and Physiological Effects of Visual Sweeps Training Exercise, 2-Arm Model
Brief Title: Behavioral and Physiological Effects of Visual Training
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RES-203-2007
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Healthy
Keywords: ACRD; Visual Memory; Visual Perception; Speed; Computerized; SAAGE; Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (No Intervention): No contact control (NCC)
- II (Experimental): Computerized, SAAGE-designed, visual memory-based cognitive training
  Interventions: Behavioral: SAAGE-designed, visual memory-based cognitive training

INTERVENTIONS:
Behavioral: SAAGE-designed, visual memory-based cognitive training — Training sessions take 40 minutes per day, five days per week for a total goal of 15, 40-minute sessions.
  Other Names: Hawkeye
  Arms: II

SUMMARY:
The primary objective of this study is to evaluate the learnability of a 3 week, 40 minutes per day, 5 day per week, computer-based visual training exercise by healthy mature individuals undergoing normal aging.

DETAILED DESCRIPTION:
Virtually all adults will suffer a decline in their cognitive capacities to some degree. Typically, cognitive decline is characterized by a slow, progressive decline in abilities (frequently in memory, attention, inhibition and speed of processing) relative to younger adults, commonly called normal aging, age-associated memory impairment, age-consistent memory impairment, benign senescent forgetfulness, late-life forgetfulness, ageing-associated cognitive decline, and the preferred term, age-related cognitive decline (ARCD) As virtually all adults experience a reduction in their cognitive abilities with age, ARCD has generally been considered to be a normal, inevitable, and irreversible part of aging; and the extremely severe forms of pathological cognitive decline (e.g., Alzheimer's disease, AD) have dominated therapeutic research in this area. However, ARCD represents an important cause of quality of life decline in almost every older adult, as the impact of forgetfulness and mental slowing increasingly change the abilities of individuals to successfully manage their day-to-day activities. Therapeutic approaches targeting the specific problems of ARCD in normal aging (as opposed to the pathological problems of AD) would unto themselves represent important clinical advances.

This trial investigates the effects of a computer-based visual training exercise built on the principles of positive brain plasticity and designed for use by healthy mature individuals. The program is specifically designed to improve the fidelity of sensory representations in early visual cortex.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older at the time of consent.
* Mini-Mental Status Examination (MMSE) score of 26 or higher.
* Adequate visual capacity adequate to read.
* Adequate hearing capacity.
* Willing and able to commit to study time requirements.

Exclusion Criteria:

* Self-report of current diagnosis or history of major neurological illness.
* Self-report of current diagnosis or history of psychiatric illness. c. History of psychiatric hospitalization in the past twenty years.
* History of a stroke, transient ischemic attack (TIA) or traumatic brain injury within the past year; or lifetime history of stroke, TIA, or traumatic brain injury that has left residual expressive or receptive language problems. - Fibromyalgia or symptoms of severe tremor.
* Self-report of current substance abuse, including alcoholism.
* Current useof medications with substantial CNS effects. Inappropriate behaviors during screening or baseline visits.
* Inability to perform behavioral evaluations.
* Participant is not capable of giving informed consent or unable to comprehend and/or follow instructions.
* Participant is enrolled in a concurrent clinical study that could affect the outcome of this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-08; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
Improvement in visual memory assessment after training or no-contact period. | 6-8 weeks

SECONDARY OUTCOMES:
Improvement on at least 1 of the Computerized Visual Attention, Speed and Memory Tests conducted. | 6-8 weeks
Improvement on the computerized cognitive assessments. | 6-8 weeks
Improvement on exercise-based assessments. | 6-8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L Hardy, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco Bay Area, California, United States

REFERENCES:
- [Background] Bischkopf J, Busse A, Angermeyer MC. Mild cognitive impairment--a review of prevalence, incidence and outcome according to current approaches. Acta Psychiatr Scand. 2002 Dec;106(6):403-14. doi: 10.1034/j.1600-0447.2002.01417.x. PMID 12392483
- [Background] Fillit HM, Butler RN, O'Connell AW, Albert MS, Birren JE, Cotman CW, Greenough WT, Gold PE, Kramer AF, Kuller LH, Perls TT, Sahagan BG, Tully T. Achieving and maintaining cognitive vitality with aging. Mayo Clin Proc. 2002 Jul;77(7):681-96. doi: 10.4065/77.7.681. PMID 12108606
- [Background] Ahissar E, Nagarajan S, Ahissar M, Protopapas A, Mahncke H, Merzenich MM. Speech comprehension is correlated with temporal response patterns recorded from auditory cortex. Proc Natl Acad Sci U S A. 2001 Nov 6;98(23):13367-72. doi: 10.1073/pnas.201400998. PMID 11698688
- [Background] Park HL, O'Connell JE, Thomson RG. A systematic review of cognitive decline in the general elderly population. Int J Geriatr Psychiatry. 2003 Dec;18(12):1121-34. doi: 10.1002/gps.1023. PMID 14677145
- [Background] Scarmeas N, Stern Y. Cognitive reserve: implications for diagnosis and prevention of Alzheimer's disease. Curr Neurol Neurosci Rep. 2004 Sep;4(5):374-80. doi: 10.1007/s11910-004-0084-7. PMID 15324603
- See also: Click here for more information about computerized cognitive training — http://www.positscience.com